CLINICAL TRIAL: NCT03743948
Title: Non Invasive Prenatal Diagnosis on Isolated Circulating Fetal Trophoblastic Cells (CFTC) for Monogenic Diseases
Brief Title: NIPD of CFTC by WGA Coupled to Mini-exome Sequencing
Acronym: DIAFEXOME
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University Hospital, Montpellier (Other)
Collaborators: ABM Industries (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: RECHMPL18_0281
Record Dates: First submitted 2018-11-08; First posted 2018-11-16 (Actual); Last update posted 2019-09-27 (Actual); Status verified 2018-11

CONDITIONS: Monogenic Diseases
Keywords: Non Invasive Prenatal Diagnosis; Circulating Fetal Trophoblastic Cells; monogenic disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Expectant couple at risk of transmitting a monogenic disease. (Experimental): Expectant couple (pregnant woman from 9 weeks of gestation and spouse) at risk of transmitting a monogenic disease among the genes included in the trusight one expanded sequencing kit (Illumina).
  Interventions: Genetic: Non invasive prenatal diagnosis

INTERVENTIONS:
Genetic: Non invasive prenatal diagnosis — 15 pregnant women and their spouses Search for the familial mutation on isolated circulating fetal trophoblastic cells from maternal blood

SUMMARY:
The purprose of this study is to develop a single test based on circulating fetal trophoblastic cells (CFTC) analysis from maternal blood, searching for the familial mutation for a wide range of monogenic diseases.

DETAILED DESCRIPTION:
Context:

Non Invasive Prenatal Diagnosis (NIPD), based on the analysis of circulating cell-free fetal DNA (cff-DNA) is very promising for early diagnosis of monogenic diseases. Such an approach is a safer alternative to invasive methods of prenatal testing (amniocentesis or choriocentesis) which entails a significant risk of miscarriage (0.5%-1%). However, technical issues related to the characteristics of cff-DNA remain, and NIPD techniques require long process development which are specific for a gene and/or a particular mutation.

Objectives:

The objective of this study is to complete our offer of NIPD by developing an approach on isolated Circulating Trophoblastic Fetal Cells (CFTC) adapted to the analysis of the genes and mutations involved in current prenatal testing requests.

Methodology :

The blood of pregnant women from 9 weeks of gestation for which a prenatal testing is requested will be collected.

CFTC isolation using Circulating Tumor Cells (CTCs) enrichment systems will be followed by whole genome amplification coupled to mini-exome sequencing and bioinformatic filtering that will be specific to the prenatal testing indication.

The study will be carried out in 2 stages:

* analytical validation of the method by studying the data quality of the sequencing of targeted genes that are frequently subject to prenatal testing (see prenatal testing diseases list from "ABM DPN 2014" in Appendix 2).
* clinical evaluation of the method by checking the concordance between the results obtained by our new approach versus those obtained by standard procedure (amniocentesis or choriocentesis) for 15 pregnant women.

Expected results and perspectives:

The purpose of this study is to establish the proof of concept of a semi-universal NIPD method based on a simple maternal blood test that could be applied on most rare diseases requiring prenatal testing.

This NIPD approach would reduce the number of invasive procedures and thus eliminate the risk of miscarriage due to amniocentesis or choriocentesis. It would also enable national access to this NIPD test for a wide range of rare diseases.

ELIGIBILITY:
Inclusion Criteria:

* older than 18 years old
* pregnant woman between 9 and 34 weeks of gestation
* Couple undergoing prenatal diagnosis for a monogenic disease caused by point mutation(s)
* Written informed consent was obtained for the study
* Prenatal diagnosis has been programmed for the current pregnancy during which maternal blood is collected
* Couple molecular diagnosis results for a monogenic disease caused by point mutation(s) MUST BE AVAILABLE.

Exclusion criteria:

* Couple Genomic DNA are unavailable
* Subjects at risk of transmitting the family disease, but not wishing to know their molecular status
* Individuals under guardianship by court order

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2018-12-19 (Actual); Primary Completion 2019-08-27 (Actual); Study Completion 2019-12-30 (Estimated)

PRIMARY OUTCOMES:
Concordance rate between cell-based genetic non invasive prenatal test and gold standard prenatal test (choriocentesis or amniocentesis). | at 36 month
  Analysis of the concordance of the prenatal results obtained by our new NIPD (Non-Invasive Prenatal Diagnosis) approach and those blindly obtained during the gold-standard prenatal genetic test will be carried out for each pregnant woman participating in the study.

SECONDARY OUTCOMES:
Non Invasive Prenatal Diagnostic test failure rate. | at 36 month
  Count of the women enrolled for whom NIPD test will be inconclusive (because of insufficient circulating fetal cells isolation or allele drop out making accurate genotyping impossible).

CONTACTS AND LOCATIONS:
Overall Officials: Claire Guissart, PhD-PharmD, Principal Investigator — molecular genetics
Locations (1):
- INSERM-Hospital,, Montpellier, Herault, France

IPD SHARING:
Plan to Share IPD: No